CLINICAL TRIAL: NCT00249964
Title: Phase I Dose Finding Clinical Trial of Combination Paclitaxel, Carboplatin and Temozolomide for Subjects With Solid Tumor Malignancies.
Brief Title: Combination Paclitaxel, Carboplatin and Temozolomide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0100C
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Lung Diseases; Cancer
Keywords: Extensive or recurrent small cell lung cancer Phase I; Paclitaxel, Carboplatin, Temozolomide
MeSH Terms: conditions — Lung Diseases; Neoplasms | interventions — Carboplatin; Paclitaxel; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Treatment (Experimental): Paclitaxel at 175 mg/m2 + Carboplatin at area under the curve (AUC) 5 on day 1. Then, Temozolomide at the doses described under "Interventions" from day 2 to day 6 (a total of 5 days).
  Cycle length is 21 days.
  Interventions: Drug: Combination Treatment - Cohort 1; Drug: Combination Treatment - Cohort 2; Drug: Combination Treatment - Cohort 3; Drug: Combination Treatment - Cohort 4

INTERVENTIONS:
Drug: Combination Treatment - Cohort 1 — Paclitaxel at 175 mg/m2 intravenously + Carboplatin at AUC 5 intravenously on day 1.
  Temozolomide at 75 mg/m2 per day from day 2 to day 6.
  Other Names: Paraplatin (Carboplatin); Taxol (Paclitaxel); Temodar (Temozolomide)
Drug: Combination Treatment - Cohort 2 — Paclitaxel at 175 mg/m2 intravenously + Carboplatin at AUC 5 intravenously on day 1.
  Temozolomide at 100 mg/m2 per day from day 2 to day 6.
  Other Names: Paraplatin (Carboplatin); Taxol (Paclitaxel); Temodar (Temozolomide)
Drug: Combination Treatment - Cohort 3 — Paclitaxel at 175 mg/m2 intravenously + Carboplatin at AUC 5 intravenously on day 1.
  Temozolomide at 125 mg/m2 per day from day 2 to day 6.
  Other Names: Paraplatin (Carboplatin); Taxol (Paclitaxel); Temodar (Temozolomide)
Drug: Combination Treatment - Cohort 4 — Paclitaxel at 175 mg/m2 intravenously + Carboplatin at AUC 5 intravenously on day 1.
  Temozolomide at 150 mg/m2 per day from day 2 to day 6.
  Other Names: Paraplatin (Carboplatin); Taxol (Paclitaxel); Temodar (Temozolomide)

SUMMARY:
The purpose of this study is to determine the maximum tolerable dose of temozolomide in combination with fixed dose of paclitaxel and carboplatin and to determine the overall tumor response rate with this combination and to determine the duration of response.

DETAILED DESCRIPTION:
The objective of the research study is to test a combination of drugs to treat small cell lung cancer which has spread beyond the lungs (extensive cancer) or come back after earlier treatment (recurrent cancer).

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Karnofsky performance status (KPS) of greater than or equal to 70 (Appendix B)
3. Laboratory values (performed within 14 days prior to study drug administration, inclusive).

   1. Absolute neutrophil count (ANC) >1500/mm3
   2. Platelet count >100,000/mm3
   3. Hemoglobin >10 g/dl or 100 g/l
   4. BUN and serum creatinine <1.5 times upper limit of laboratory normal
   5. Total and direct bilirubin <1.5 times upper limit of laboratory normal
   6. SGOT and SGPT <3 times upper limit of laboratory normal
   7. Alkaline Phosphatase <3 times upper limit of laboratory normal
4. A life expectancy of greater than 12 weeks
5. Subjects must give written informed consent.
6. Biopsy proven small cell lung cancer.
7. CT of chest, abdomen, pelvis and MRI of head
8. Patients with brain metastases should be asymptomatic to enter the study

Exclusion Criteria:

1. No recovery from all active toxicities of prior therapies.
2. Subjects who are poor medical risks because of non-malignant systemic disease as well as those with acute infection treated with intravenous antibiotics.
3. Frequent vomiting or medical condition that could interfere with oral medication intake (eg, partial bowel obstruction).
4. Concurrent malignancies at other sites with the exception of surgically cured carcinoma in-site of the cervix and basal or squamous cell carcinoma of the skin. Prior malignancies which have not required anti-tumor treatment within the preceding 24 months are eligible.
5. Known HIV positivity or AIDS-related illness.
6. Pregnant or nursing women.
7. Women of childbearing potential who are not using an effective method of contraception. Women of childbearing potential must have a negative serum pregnancy test 24 hours prior to administration of study drug and be practicing medically approved contraceptive precautions.
8. Men who are not advised to use an effective method of contraception.
9. Progression of disease on prior chemotherapy with paclitaxel and carboplatin, either as single agent or in combination.
10. Known hypersensitivity reaction to taxoid or platinum compound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Temozolomide in Combination with Fixed Doses of Paclitaxel and Carboplatin | 4 months
  Temozolomide was administered at different dose levels (see Cohorts 1-4) until the maximum tolerated dose (MTD) was reached. MTD is the dose at which 0/6 or 1/6 patients in the cohort experience dose limiting toxicity (DLT) during the first 4 week cycle with the next higher dose having at least 2/3 or 2/6 patients experiencing DLT. DLT will have occurred when the patient has 1 or more Grade 4 hematologic or nonhematologic toxicities. A DLT must occur in the first cycle of the combination and must be at least possibly attributed to the treatment regimen. Toxicities will be graded according to the NCI CTCAE Version 3.0.

SECONDARY OUTCOMES:
Tumor response rate | 7 months
  Tumor response is evaluated according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0 as determined by the investigator. Complete response (CR): Disappearance of all evidence of target and non-target lesions. Partial response (P): >= 30% reduction from baseline in the sum of the longest diameter of all lesions. CR and PR criteria should be met again after 4 weeks and before 6 weeks after initial assessment. Stable Disease (SD): Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. Progressive disease (PD) for target lesions: >= 20% increase in the sum of diameters of the target lesions taking as reference the smallest sum on study, and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered . PD for non-target lesions is defined as unequivocal appearance of one or more new malignant lesions or unequivocal progression of existing non-target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States